CLINICAL TRIAL: NCT04109612
Title: Improving Stroke Care in Greece in Terms of Management, Costs and Health Outcomes- Stroke Units Necessity for Patients (SUN4P)
Brief Title: Improving Stroke Care in Greece in Terms of Management, Costs and Health Outcomes-
Acronym: SUN4P
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Hellenic Foundation for Research and Innovation (Unknown); General Secretariat for Research and Technology (Unknown); Hellenic Stroke Organization (Unknown)
Responsible Party: Principal Investigator, OLGA SISKOU, Senior Researcher, National and Kapodistrian University of Athens
Other Study IDs: 15117
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Cerebrovascular Disorders
Keywords: stroke; stroke care; stroke units; value of stroke care
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objectives of the proposed project are:

1. To provide essential data on acute stroke management (quality indicators) incorporating hard clinical outcomes that will contribute to an ongoing process of quality improvement
2. To develop an interactive multichannel platform, for collecting, cleansing and curating high quality in-hospital and follow up data, applying multidimensional quality assessment analysis, providing statistical and analytic reports, monitoring behavioral changes and supporting overall project's management.
3. To evaluate patients' and physicians' experiences and their impact on stroke management.
4. To assess severe negative impact of stroke on the life of survivors including quality of life and disability
5. To measure health related and non- health (loss of productivity, informal care) related national expenditure for stroke care using a bottom up approach
6. To evaluate the value of care focusing on health outcomes compared with total costs of achieving them

DETAILED DESCRIPTION:
A prospective cohort multicenter study of patients with first ever acute stroke, hemorrhagic and ischemic, (ICD-10 codes: I61, I63 and I64) admitted within 48 hours of symptoms onset to seven NHS and University hospitals will be conducted. About 1,000 patients (2% of all new cases/annually) will be recruited from six urban and semi-urban areas with 5.5 mil people (50% of Greek population), reporting 25,000 discharged stroke cases annually (53% of all stroke discharges), according to data derived from Hellenic Statistical Authority. All patients will be followed for three months. Moreover, a sub-group of the 300 firstly recruited patients will be followed for a year to obtain data on post hospital health and social needs, health services utilization (medication, rehabilitation, outpatient visits) and productivity loss . Patient enrolment and follow up is estimated to last 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemorrhagic or ischemic stroke (ICD-10: I61, I63 and I64)
* Patients with First ever acute stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 1,000 first ever stroke patients (2% of all new cases/annually) will be recruited from six urban and semi-urban areas with 5.5 mil people (50% of Greek population), reporting 25,000 discharged stroke cases annually. All patients will be followed for three months.
Sampling Method: Non-Probability Sample
Enrollment: 913 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Mortality | Through hospitalization completion, an average of 10 days
  Patient based stroke (inpatient and outpatient) mortality
Mortality | One month
  Patient based stroke (inpatient and outpatient) mortality
Mortality | Three months
  Patient based stroke (inpatient and outpatient) mortality
Modified Rankin Scale (mRS) score | Through hospitalization completion, an average of 10 days
  mRS measures the degree of disability or dependence in the daily activities of patients after a stroke or other causes of neurological disability (0: no symptoms at all - 6: Dead)
Modified Rankin Scale (mRS) score | One month
  mRS measures the degree of disability or dependence in the daily activities of patients after a stroke or other causes of neurological disability (0: no symptoms at all - 6: Dead)
Modified Rankin Scale (mRS) score | Three months
  mRS measures the degree of disability or dependence in the daily activities of patients after a stroke or other causes of neurological disability (0: no symptoms at all - 6: Dead)
National Institutes of Health Stroke Scale (NIHSS) score | Through hospitalization completion, an average of 10 days
  NIHSS is a method for assessing the severity of a stroke experienced by a patient (0: No Stroke Symptoms, 42:Severe Stroke)
National Institutes of Health Stroke Scale (NIHSS) score | One month
  NIHSS is a method for assessing the severity of a stroke experienced by a patient (0: No Stroke Symptoms, 42: Severe Stroke)
National Institutes of Health Stroke Scale (NIHSS) score | Three months
  NIHSS is a method for assessing the severity of a stroke experienced by a patient (0: No Stroke Symptoms, 42: Severe Stroke)
Cost | Through hospitalization completion, an average of 10 days
  Average cost per patient
Cost | One month
  Average cost per patient
Cost | Three months
  Average cost per patient

CONTACTS AND LOCATIONS:
Overall Officials: OLGA SISKOU, PhD, Principal Investigator — Senior Researcher on Health and Nursing Economics and Management; GEORGE NTAIOS, PhD, Principal Investigator — Head of Physicians /Nurses Team; GEORGE PAPASTEFANATOS, PhD, Principal Investigator — Head of IT Team
Locations (10):
- Greece (10):
  - National and Kapodistrian University of Athens, Athens
  - Aiginiteio Hospital of Athens, Athens
  - General Hospital of Athens Alexandra, Athens
  - Hellenic Stroke Organization, Athens
  - Laiko General Hospital of Athens, Athens
  - Chania General Hospital St George, Chania
  - University General Hospital of Ioannina, Ioannina
  - General University Hospital of Larisa, Larissa
  - University General Hospital of Thessaloniki Ahepa, Thessaloniki
  - General Hospital of Tripoli Evaggelistria, Tripoli

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Project site — http://www.sun4patients.gr/en
- See also: Paper entitled:Access of Stroke Patients' to Optimal Healthcare Technology in Greece: Messages to Policy Makers — https://pubmed.ncbi.nlm.nih.gov/32604692
- See also: Paper entitled: Developing Patients' Experiences Database After Hospital Discharge: Another Step In Improving Stroke Care — https://pubmed.ncbi.nlm.nih.gov/32604697
- See also: Paper entitled: Sun4Patients Web Platform: Facilitating Long-Term Monitoring of Stroke Patients — https://pubmed.ncbi.nlm.nih.gov/32604689/
- See also: Paper entitled: Stroke Units Necessity for Patients, Web-Based "SUN4P" Registry: Descriptive Characteristics of the Population — https://pubmed.ncbi.nlm.nih.gov/35062158/
- See also: Paper entitled:Assessing Staff's and Stroke Patients' Experiences in 8 Hospitals in Greece: Results from a Prospective Multi-Center Study ("SUN4Patients") — https://pubmed.ncbi.nlm.nih.gov/35062174/
- See also: Paper entitled: Inpatient Cost of Stroke Care in Greece: Preliminary Results of the Web-Based "SUN4P" Registry — https://pubmed.ncbi.nlm.nih.gov/35062185/